CLINICAL TRIAL: NCT02530489
Title: Triple-Negative First-Line Study: Neoadjuvant Trial of Nab-Paclitaxel and MPDL3280A, a PDL-1 Inhibitor in Patients With Triple Negative Breast Cancer
Brief Title: Nab-Paclitaxel and Atezolizumab Before Surgery in Treating Patients With Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1043; NCI-2015-01537 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-1043 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Breast Adenocarcinoma; Invasive Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (atezolizumab, nab-paclitaxel) (Experimental): NEOADJUVANT: Patients receive atezolizumab IV over 60 minutes on day 1 and nab-paclitaxel IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  SURGERY: Patients undergo definitive breast surgery within 6 weeks of the completion of treatment.
  ADJUVANT: Within 4 weeks after surgery, patients receive atezolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel

SUMMARY:
This phase II trial studies how well nab-paclitaxel and atezolizumab before surgery work in treating patients with triple negative breast cancer (breast cancer cells that do not have estrogen receptors, progesterone receptors, or large amounts of human epidermal growth factor receptor 2 protein). Drugs used in chemotherapy, such as nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving nab-paclitaxel and atezolizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. This drug combination before surgery may be an effective treatment for triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the rate of pathologic complete response (pCR)/residual cancer burden (RCB)-0 + residual cancer burden (RCB)-I responses in patients with triple negative breast cancer (TNBC), who were non-responders to initial anthracycline and cyclophosphamide chemotherapy, treated with atezolizumab in combination with nab-paclitaxel in the neoadjuvant setting.

SECONDARY OBJECTIVES:

I. To estimate progression free survival (PFS) distribution of triple negative breast cancer (TNBC) patients who were non-responders to initial anthracycline and cyclophosphamide chemotherapy, treated with atezolizumab in combination with nab-paclitaxel in the neoadjuvant setting.

II. To determine the safety of atezolizumab in combination with nab-paclitaxel in the neoadjuvant setting.

EXPLORATORY OBJECTIVE:

I. To investigate the association between biomarkers in the peripheral blood and tumor tissue with efficacy for TNBC patients treated with atezolizumab in combination with nab-paclitaxel in the neoadjuvant setting.

OUTLINE:

NEOADJUVANT: Patients receive atezolizumab intravenously (IV) over 60 minutes on day 1 and nab-paclitaxel IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

SURGERY: Patients undergo definitive breast surgery within 6 weeks of the completion of treatment.

ADJUVANT: Within 4 weeks after surgery, patients receive atezolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically confirmed primary invasive adenocarcinoma of the breast with the size of the primary tumor being at least 1.5 cm, or at least 1 biopsy confirmed involved lymph node > 1.5 cm, on imaging by either mammography, ultrasound or breast magnetic resonance imaging (MRI)
* Estrogen receptor (ER) and progesterone receptor (PR) expression both < 10% by immunohistochemistry (IHC) and human epidermal growth factor receptor 2 (HER2) negative or non-amplified as determined by the current American Society of Clinical Oncology (ASCO)-College of American Pathologists (CAP) criteria which are as follows: HER2 testing by IHC as 0 or 1+; if HER2 is 2+, ISH (in situ hybridization) must be performed; HER2 is positive for gene amplification if: - IHC 3+ based on circumferential membrane staining that is complete, intense - ISH positive based on:

  * Single-probe average HER2 copy number >= 6.0 signals/cell
  * Dual-probe HER2/chromosome enumeration probe (CEP)17 ratio >= 2.0; with an average HER2 copy number >= 4.0 signals/cell
  * Dual-probe HER2/CEP17 ratio >= 2.0; with an average HER2 copy number < 4.0 signals/cell
  * Dual-probe HER2/CEP17 ratio < 2.0; with an average HER2 copy number >= 6.0 signals/cell
* No prior treatment for primary invasive adenocarcinoma of the breast such as irradiation, chemotherapy, hormonal therapy, immunotherapy, investigational therapy or surgery other than the anthracycline and cyclophosphamide chemotherapy with or without 5-fluorouracil; treatment for ductal carcinoma in situ is allowed, such as surgery, hormonal therapy and radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Baseline multi gated acquisition scan (MUGA) or echocardiogram scans with left ventricular ejection fraction (LVEF) of > 50%
* Absolute neutrophil count (ANC) >= 1500 cells/uL
* White blood cell counts (WBC) > 2500/uL
* Lymphocyte count >= 300/uL
* Platelet count >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) with the following exception: patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN; this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 6 months after the last dose of investigational product in such a manner that the risk of pregnancy is minimized; men on study and for at least 6 months after the last dose of nab-paclitaxel also must be using contraception; women of childbearing potential (WOCBP) are women who have not been postmenopausal greater than 1 year or undergone a hysterectomy and/or bilateral oophorectomy
* Negative serum or urine pregnancy test for women within 72 hours of receiving the first dose of the study medication for women of childbearing potential
* Classified as having insufficient tumor shrinkage by imaging (< 80% shrinkage after 4 cycles of anthracycline-based chemotherapy based upon diagnostic imaging)

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Known metastatic disease
* Disease free of prior malignancy for < 5 years with the exception of curatively treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, or transitional cell carcinoma
* Has received prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), anti-programmed cell death ligand 2 (PD-L2), anti-cluster of differentiation (CD)137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has had major surgery within 21 days before cycle 1, day 1
* Uncontrolled inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Serious intercurrent infections or non-malignant medical illness that are uncontrolled or the control of which may be jeopardized by this therapy
* Psychiatric disorders or other conditions rendering the subject incapable of complying with the requirements of the protocols
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis; patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible; patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible; patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions: patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations, rash must cover less than 10% of body surface area (BSA), disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%), no acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Known to be human immunodeficiency virus positive
* Patients with prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C; patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti HBc] antibody test) are eligible; patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study; influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug, whichever is shorter
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents), or anticipated requirement for systemic immunosuppressive medications during the trial; patients who have received acute, low dose, systemic immunosuppressant medications (e.g., dexamethasone prior to the anthracycline-based chemotherapy for nausea) may be enrolled in the study; the use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed
* Concurrent disease or condition that would interfere with study participation or safety, such as any of the following:

  * Active, clinically significant infection either grade > 2 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 or requiring the use of parenteral anti-microbial agents within 14 days before day 1 of study drug
  * Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders
  * Non-healing wound, ulcer, or bone fracture
* Known hypersensitivity to any of the components of atezolizumab or nab-paclitaxel
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR)/residual cancer burden (RCB)-0 + RCB-I responses in patients with triple-negative breast cancer | Up to 3 years
  The proportion of patients with pCR (RCB-0) or RCB-I will be estimated as the response rate along with an appropriate 95% confidence interval. The proportion of patients in the remaining RCB categories will be estimated with confidence intervals as well.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From the date of enrollment until the date of progression or death without evidence of progression, assessed up to 3 years
  The PFS distribution will be estimated using the Kaplan-Meier method.
Overall survival (OS) | Up to 3 years
  The OS distribution will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Yam, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yam C, Mittendorf EA, Garber HR, Sun R, Damodaran S, Murthy RK, Ramirez D, Karuturi M, Layman RM, Ibrahim N, Rauch GM, Adrada BE, Candelaria RP, White JB, Ravenberg E, Clayborn A, Ding QQ, Symmans WF, Prabhakaran S, Thompson AM, Valero V, Tripathy D, Huo L, Moulder SL, Litton JK. A phase II study of neoadjuvant atezolizumab and nab-paclitaxel in patients with anthracycline-resistant early-stage triple-negative breast cancer. Breast Cancer Res Treat. 2023 Jun;199(3):457-469. doi: 10.1007/s10549-023-06929-9. Epub 2023 Apr 15. PMID 37061619
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT02530489/ICF_000.pdf